CLINICAL TRIAL: NCT02890589
Title: Strut Coverage With SYNERGY Stents and Bioresorbable Vascular Scaffold in Acute Myocardial Infarction: An Intracoronary Optical Coherence Tomography Randomized Study
Brief Title: Strut Coverage With SYNERGY Stents and Bioresorbable Vascular Scaffold in Acute Myocardial Infarction
Acronym: COVER-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/15/7743
Record Dates: First submitted 2016-06-28; First posted 2016-09-07 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2019-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; ST (Software Test) -elevation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYNERGY Stent (Experimental): The SYNERGY™ stent is a Device marked CE (European Conformity), platinum chromium coronary stent, currently developped by Boston Scientific™. This stent has been designed with the goal of providing optimal and rapid healing within the vessel using a bioabsorbable polymer to elute everolimus.
  Interventions: Device: SYNERGY stent
- BVS device (Experimental): The ABSORB Everolimus-eluting Bioresorbable Vascular Scaffold (BVS 1.1, Abbott Vascular, California, USA, CE approved) is Device marked CE, currently the most studied PLA (Polylactic acid) based scaffold. It consists of PLLA (Poly I-lactic acid) backbone with 1:1 PDLLA (Poly-DL Lactic Acid) drug surface coating and a total strut thickness of 156 μm.
  Interventions: Device: ABSORB (Everolimus-eluting Bioresorbable Vascular Scaffold)

INTERVENTIONS:
Device: SYNERGY stent — Coronary angiography will assess the presence of at least one eligible coronary lesion requiring stent implantation before revascularization by angioplasty.
  Stent will be implanted according to manufacturer's and competent authority recommendations.
  Other Names: SYNERGY (Platinum chromium coronary stent)
  Arms: SYNERGY Stent
Device: ABSORB (Everolimus-eluting Bioresorbable Vascular Scaffold) — Coronary angiography will assess the presence of at least one eligible coronary lesion requiring stent implantation before revascularization by angioplasty.
  Stent will be implanted according to manufacturer's and competent authority recommendations.
  Other Names: ABSORB
  Arms: BVS device

SUMMARY:
To assess strut coverage in patients presenting an acute myocardial infarction and treated either with the SYNERGY stent or the Bioresorbable Vascular Scaffold, through a parallel group design.

DETAILED DESCRIPTION:
Single center, simple-blind randomized controlled trial, comparing the SYNERGY stent with the BVS device through a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome with ST-elevation,
* One culprit lesion eligible for percutaneous coronary intervention (PCI) with stent implantation,
* Reference vessel measuring 2.5 mm to 3.75 mm per visual estimation, without extreme vessel tortuosity,
* thrombolysis in myocardial infarction (TIMI) 3 flow before stent deployment in the target vessel,
* Patient with at least 1 lesion eligible for planned PCI next to the culprit lesion,
* Patient affiliated to the French national health care system,
* Patient agreed to participate after full information on the study (signature of an informed consent).

Exclusion Criteria:

* Acute coronary syndrome with ST-elevation,
* One culprit lesion eligible for percutaneous coronary intervention (PCI) with stent implantation,
* Reference vessel measuring 2.5 mm to 3.75 mm per visual estimation, without extreme vessel tortuosity,
* TIMI 3 flow before stent deployment in the target vessel,
* Patient with at least 1 lesion eligible for planned PCI next to the culprit lesion,
* Patient affiliated to the French national health care system,
* Patient agreed to participate after full information on the study (signature of an informed consent).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of uncovered stent struts at 3-months | at 3-months
  To assess strut coverage

SECONDARY OUTCOMES:
Percentage of malposed uncovered struts | at 3 months
  Assessed by optical coherence tomography
Frequency of abnormal intrastent tissue | at 3 months
  Assessed by optical coherence tomography
Percentage of net volume obstruction | at 3 months
  Assessed by optical coherence tomography
Rates of in-stent late loss | at 3 months
Rates of in-segment late loss | at 3 months
Rates of binary restenosis | at 3 months
Plasma CXCL10 protein as a potential of re-endothelialization | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Didier CARRIE, MD Phd, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Didier CARRIE, Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lhermusier T, Ohayon P, Boudou N, Bouisset F, Campelo-Parada F, Roncalli J, Elbaz M, Carrie D. Re-endothelialisation after Synergy stent and Absorb bioresorbable vascular scaffold implantation in acute myocardial infarction: COVER-AMI study. Trials. 2019 Apr 11;20(1):210. doi: 10.1186/s13063-019-3293-8. PMID 30975219